CLINICAL TRIAL: NCT02308176
Title: Effectiveness of a Mobile Application as an Adjunct to Medical Advice to Promote Healthy Habits (Diet and Sport) in a Population of Patients Obese or Overweight Adults Patients
Brief Title: Effectiveness of a Mobile Application as an Adjunct to Medical Advice to Promote Healthy Habits
Acronym: AD01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Antxon Apiñaniz Fernández de LArrinoa, MAIN RESEARCHER, Basque Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AKTIDIET
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention group (Experimental): health advice and app installation in patient's mobile
  Interventions: Behavioral: APP + health advice
- control group (Placebo Comparator): health advice
  Interventions: Behavioral: health advice

INTERVENTIONS:
Behavioral: APP + health advice — health advice and reinforcement to it
  Arms: intervention group
Behavioral: health advice — health advice
  Arms: control group

SUMMARY:
INTRODUCTION: Obesity is the most common metabolic problem and its genesis and maintenance there is always a positive energy balance, with less energy expenditure than that obtained from the intake. Low physical activity is often an important factor in this lower spending. Medical advice is useful for determining changes in the habits of life of patients, however, the changes produced by the council do not last over time, so it would be necessary to establish enforcement mechanisms as with mobile technology, because it could improve the adhesion of obese patients to therapy. OBJECTIVE: Primary: To evaluate the effectiveness of an app as an adjunct to medical advice to promote healthy living habits (sport and diet) to lose weight in a population of obese or overweight adult patients. MATERIAL AND METHODS: Open randomized controlled clinical trial with clinical practice (health advice for physical activity and sport). STUDY POPULATION: Obese or overweight adults patients of Araba aged between 18-45 years who be in Contemplation stage with smartphone. Variables: Primary endpoint: Weight (kg); Secondary variables: BMI (kg/cm2); blood pressure (mm Hg); heart rate; Plasma cholesterol (mg / dl); HbA1c; score on the satisfaction questionnaire; index of physical exercise (IPAQ) (METs); quitting tobacco (yes / no); Waist circumference (cm). Statistical analysis: The primary endpoint (weight reduction) will be evaluated by covariance analysis adjusting by baseline weight, and other confounding variables (sex, age, level of education..) Simple size: 48 patients by arm plus 20% to cover losses to follow.

ELIGIBILITY:
Inclusion Criteria:

* BMI> = 25 mg / kg
* Holder smartphone
* Sign informed consent

Exclusion Criteria:

* Presence of physical or mental illnesses that prevent the realization of physical activity
* Be participating in another research project
* Pregnancy or lactation
* Patients who are on diet or drug treatment for weight loss
* History of myocardial infarction or stroke

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2015-09; Primary Completion 2017-05 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
weight reduction | at 6 months
  reduction of weight

SECONDARY OUTCOMES:
BMI | at 6 and 12 months
blood pressure | at 6 and 12 months
heart rate | at 6 and 12 months
smoking cessation | at 6 and 12 months
  quitting tobacco (yes / no)
waist circumference | at 6 and 12 months
plasma cholesterol | at 12 months
satisfaction | at 12 months
  satisfaction questionnaire
index of physical exercise | at 12 months
  index of physical exercise (IPAQ) (METs)

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Comarca Araba (Salburua Health Center), Vitoria-Gasteiz, Alava
  - Comarca Araba (Lakubizkarra Health Center), Vitoria-Gasteiz, Alava
  - Comarca Araba (Zabalgana Health Center), Vitoria-Gasteiz, Alava

REFERENCES:
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882
- [Derived] Apinaniz A, Cobos-Campos R, Saez de Lafuente-Morinigo A, Parraza N, Aizpuru F, Perez I, Goicoechea E, Trapaga N, Garcia L. Effectiveness of randomized controlled trial of a mobile app to promote healthy lifestyle in obese and overweight patients. Fam Pract. 2019 Nov 18;36(6):699-705. doi: 10.1093/fampra/cmz020. PMID 31093681